CLINICAL TRIAL: NCT06496321
Title: Morbidity of Conventional and No-touch Saphenectomy in Coronary Artery Bypass Grafting, a Randomized Non-inferiority Clinical Trial
Brief Title: Morbidity of Conventional and No-touch Saphenectomy in Coronary Artery Bypass Grafting.
Acronym: TNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cirugia Cardiaca, Uruguay (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNT
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Saphenectomy; No Touch; Coronary Artery Disease; Cardiovascular Diseases; Wound Complication
Keywords: Saphenectomy; No Touch; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Corresponds to a single-center, open, non-inferiority, randomized controlled clinical trial.
  A probability of complication of saphenectomy by conventional or "control" technique of 10% was assumed, based on studies from our institution, and according to preliminary studies we expect to find 50% more in the "no touch" technique, therefore 15%. The non-inferiority limit will be 20%. With these values, assuming a 95% confidence interval and a power (1 - beta) of 80%, and taking into account a probable 20% of lost patients, we can calculate the necessary population sample size, which was in total 52 patients; 26 people in the group with conventional technique and 26 in the "no touch".
Who Masked: Participant, Investigator
Masking Description: The patient will not know which group he was assigned to, and the researcher who will evaluate the patients postoperatively will not know either, only the surgeon at the time of performing block randomization prior to surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Experimental): 26 patients will be randomized to this group. The vein harvest technique will be the conventional one.
  Interventions: Procedure: Conventional Saphenous vein harvest
- No Touch (Experimental): 26 patients will be randomized to this group. The vein harvest technique will be the "no touch".
  Interventions: Procedure: No touch Saphenous vein harvest

INTERVENTIONS:
Procedure: Conventional Saphenous vein harvest — The conventional one involves harvesting only the vein, without perivascular tissue or the nerve.
  Other Names: Conventional Saphenectomy
  Arms: Conventional
Procedure: No touch Saphenous vein harvest — During the extraction of the saphenous vein using the "no touch" technique, it is sectioned with the perivascular adipose tissue and the saphenous nerve of the leg.
  Other Names: No touch Saphenectomy
  Arms: No Touch

SUMMARY:
A clinical research project will be carried out that will consist of a non-inferiority study. The objective is to compare the morbidity of two different surgical techniques for the extraction of the internal saphenous vein, intended to be used as a conduit in coronary bypass.

DETAILED DESCRIPTION:
Current clinical trials have shown that the no-touch saphenectomy technique has had a positive impact on the short- and long-term patency of coronary bypass, compared to the conventional extraction technique. It is important to highlight that the conventional technique is the most used in our country (Uruguay, South America), while the "no touch" has fallen into disuse.

Given this disparity in the application of the techniques, it is considered essential to compare both methods in terms of morbidity. For this purpose, a prospective randomized clinical trial will be carried out.

The primary objective is to demonstrate the non-inferiority of the "no touch" technique over the conventional technique in terms of wound morbidity in patients undergoing coronary revascularization, within a non-inferiority margin. Defining morbidity as the combined result of local infection, hematoma, blisters, secretions, necrosis, wound dehiscence, paresthesias, pain and functional impotence.

The investigators will seek to achieve as a specific objective the incidence of each of the study factors: local infection, hematoma, blisters, secretions, necrosis, wound dehiscence, paresthesias, pain, functional impotence and then compare them between both groups at different times.

The anatomopathological study of some of the saphenous vein preparations, one "no touch" and the other conventional, will also be carried out using optical microscopy and ultrastructural comparisons using transmission electron microscopy.

Additionally, patients will be offered computed tomography angiography every year to evaluate graft patency.

There are not many relevant randomized clinical trials that compare the morbidity of this technique with the conventional one. In this context, we consider it crucial to evaluate whether there are significant differences in terms of wound morbidity in the mid-postoperative period (1 week), late (1 month) and long-term postoperative period (6 months).

We will define each variable previously: it will be considered to have a local infection when the wound shows signs of flow and it has been necessary to start antibiotic treatment, hematoma when there is a tumor or abnormal hardening caused by the accumulation of blood, flictenes when a skin blister appears on the wound that contains watery substances and not pus, secretions when the wound secretes a liquid (serous, bloody, purulent), necrosis when there is a necrotic plaque in the wound larger than 10 x 10 mm, dehiscence of the wound when the suture loses continuity, paresthesia when there is a tingling sensation due to an irritative sensitivity disorder, pain when it is located at the level of the wound and functional impotence when it prevents or limits ambulation.

Through multivariate analysis, the relationship with independent factors will be analyzed.

Null hypothesis: "no touch" saphenectomy is inferior to the conventional technique.

Alternative hypothesis: "no touch" saphenectomy is not inferior to the conventional technique.

Existing studies have focused their attention on evaluating the patency of the ducts; however, there is a lack of solid information on the morbidity associated with this technique in the lower limb of patients. Currently, the most widely used technique remains the conventional one, which involves a continuous incision in the skin of the leg or thigh. In this technique, a dissection of the subcutaneous tissue surrounding the vein is performed, the collaterals are ligated, and the free venous duct is sectioned. The length of the conduit varies depending on the amount of bypass to be performed. During the extraction of the saphenous vein using the "no touch" technique, it is sectioned with the perivascular adipose tissue and the saphenous nerve of the leg, therefore, it is of great interest for us to evaluate the incidence of the postoperative complications, previously mentioned, and compare these results with those obtained through the conventional technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coordination coronary revascularization surgery, in which it is necessary to use the internal saphenous vein as a conduit.

Exclusion Criteria:

* Emergency surgeries.
* Poor metabolic control (HbA1c > 6.5%).
* Chronic venous insufficiency or chronic obstructive arteriopathy of the lower limbs.
* Type II obesity (BMI>35).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of the "no touch" technique over the conventional technique in terms of wound morbidity. | 1 week, 1 month, 6 months
  Our primary objective will be to demonstrate the non-inferiority of the "no touch" technique over the conventional technique in terms of wound morbidity in patients undergoing coronary revascularization, within a non-inferiority margin. Defining morbidity as the combined result of local infection, hematoma, blisters, secretions, necrosis, wound dehiscence, paresthesias, pain and functional impotence.

SECONDARY OUTCOMES:
Incidence of local infection, hematoma, flictena, secretions, necrosis, wound dehiscence, paresthesia, pain, functional impotence and then compare them between both groups at different times. | 1 week, 1 month, 6 months
  Find the incidence of each of the study factors: local infection, hematoma, flictena, secretions, necrosis, wound dehiscence, paresthesia, pain, functional impotence and then compare them between both groups at different times.

OTHER OUTCOMES:
Saphenous vein bypass patency | 1 year
  Patients will be offered computed tomography angiography one year after surgery to evaluate graft patency.

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Montero, MD, Principal Investigator — Instituto Nacional de Cirugía Cardíaca
Locations (1):
- Instituto Nacional de Cirugia Cardiaca, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dashwood MR, Pinheiro BB, Souza DSR. Impact of saphenous vein harvesting on graft diameter: Supporting the no-touch technique. JTCVS Tech. 2022 Aug 18;16:105-106. doi: 10.1016/j.xjtc.2022.08.011. eCollection 2022 Dec. No abstract available. PMID 36510541
- [Result] Deb S, Singh SK, de Souza D, Chu MWA, Whitlock R, Meyer SR, Verma S, Jeppsson A, Al-Saleh A, Brady K, Rao-Melacini P, Belley-Cote EP, Tam DY, Devereaux PJ, Novick RJ, Fremes SE; SUPERIOR SVG Study Investigators. SUPERIOR SVG: no touch saphenous harvesting to improve patency following coronary bypass grafting (a multi-Centre randomized control trial, NCT01047449). J Cardiothorac Surg. 2019 May 2;14(1):85. doi: 10.1186/s13019-019-0887-x. PMID 31046806
- [Result] Gaudino M, Antoniades C, Benedetto U, Deb S, Di Franco A, Di Giammarco G, Fremes S, Glineur D, Grau J, He GW, Marinelli D, Ohmes LB, Patrono C, Puskas J, Tranbaugh R, Girardi LN, Taggart DP; ATLANTIC (Arterial Grafting International Consortium) Alliance. Mechanisms, Consequences, and Prevention of Coronary Graft Failure. Circulation. 2017 Oct 31;136(18):1749-1764. doi: 10.1161/CIRCULATIONAHA.117.027597. PMID 29084780
- [Result] Inaba Y, Yamazaki M, Ohono M, Yamashita K, Izumida H, Hayashi K, Takahashi T, Kimura N, Ito T, Shimizu H. No-touch saphenous vein graft harvesting technique for coronary artery bypass grafting. Gen Thorac Cardiovasc Surg. 2020 Mar;68(3):248-253. doi: 10.1007/s11748-019-01186-4. Epub 2019 Aug 2. PMID 31376117
- [Result] Kopjar T, Dashwood MR. Endoscopic Versus "No-Touch" Saphenous Vein Harvesting for Coronary Artery Bypass Grafting: A Trade-Off Between Wound Healing and Graft Patency. Angiology. 2016 Feb;67(2):121-32. doi: 10.1177/0003319715584126. Epub 2015 May 13. PMID 25972395
- [Result] Pettersen O, Haram PM, Winnerkvist A, Karevold A, Wahba A, Stenvik M, Wiseth R, Hegbom K, Nordhaug DO. Pedicled Vein Grafts in Coronary Surgery: Perioperative Data From a Randomized Trial. Ann Thorac Surg. 2017 Oct;104(4):1313-1317. doi: 10.1016/j.athoracsur.2017.03.076. Epub 2017 Jun 23. PMID 28648540
- [Result] Ragnarsson S, Janiec M, Modrau IS, Dreifaldt M, Ericsson A, Holmgren A, Hultkvist H, Jeppsson A, Sartipy U, Ternstrom L, Per Vikholm MD, de Souza D, James S, Thelin S. No-touch saphenous vein grafts in coronary artery surgery (SWEDEGRAFT): Rationale and design of a multicenter, prospective, registry-based randomized clinical trial. Am Heart J. 2020 Jun;224:17-24. doi: 10.1016/j.ahj.2020.03.009. Epub 2020 Mar 13. PMID 32272256
- [Result] Souza DS, Christofferson RH, Bomfim V, Filbey D. "No-touch" technique using saphenous vein harvested with its surrounding tissue for coronary artery bypass grafting maintains an intact endothelium. Scand Cardiovasc J. 1999;33(6):323-9. doi: 10.1080/14017439950141362. PMID 10622542
- [Result] Samano N, Geijer H, Liden M, Fremes S, Bodin L, Souza D. The no-touch saphenous vein for coronary artery bypass grafting maintains a patency, after 16 years, comparable to the left internal thoracic artery: A randomized trial. J Thorac Cardiovasc Surg. 2015 Oct;150(4):880-8. doi: 10.1016/j.jtcvs.2015.07.027. Epub 2015 Jul 15. PMID 26282605
- [Result] Souza DS, Dashwood MR, Tsui JC, Filbey D, Bodin L, Johansson B, Borowiec J. Improved patency in vein grafts harvested with surrounding tissue: results of a randomized study using three harvesting techniques. Ann Thorac Surg. 2002 Apr;73(4):1189-95. doi: 10.1016/s0003-4975(02)03425-2. PMID 11996262
- [Result] Souza DS, Arbeus M, Botelho Pinheiro B, Filbey D. The no-touch technique of harvesting the saphenous vein for coronary artery bypass grafting surgery. Multimed Man Cardiothorac Surg. 2009 Jan 1;2009(731):mmcts.2008.003624. doi: 10.1510/mmcts.2008.003624. PMID 24413611
- [Result] Tian M, Wang X, Sun H, Feng W, Song Y, Lu F, Wang L, Wang Y, Xu B, Wang H, Liu S, Liu Z, Chen Y, Miao Q, Su P, Yang Y, Guo S, Lu B, Sun Z, Liu K, Zhang C, Wu Y, Xu H, Zhao W, Han C, Zhou X, Wang E, Huo X, Hu S. No-Touch Versus Conventional Vein Harvesting Techniques at 12 Months After Coronary Artery Bypass Grafting Surgery: Multicenter Randomized, Controlled Trial. Circulation. 2021 Oct 5;144(14):1120-1129. doi: 10.1161/CIRCULATIONAHA.121.055525. Epub 2021 Sep 13. PMID 34510911
- [Result] Tsuneyoshi H, Setozaki S, Katayama H, Wada T, Shimomura S, Takeuchi A, Sugaya A, Komiya T. Early and Midterm Outcomes of "No-Touch" Saphenous Vein Grafts in Japanese Institutions. Braz J Cardiovasc Surg. 2022 Sep 2;37(Spec 1):42-48. doi: 10.21470/1678-9741-2022-0121. PMID 36054001
- [Result] Verma S, Lovren F, Pan Y, Yanagawa B, Deb S, Karkhanis R, Quan A, Teoh H, Feder-Elituv R, Moussa F, Souza DS, Fremes SE. Pedicled no-touch saphenous vein graft harvest limits vascular smooth muscle cell activation: the PATENT saphenous vein graft study. Eur J Cardiothorac Surg. 2014 Apr;45(4):717-25. doi: 10.1093/ejcts/ezt560. Epub 2013 Dec 9. PMID 24327455
- [Result] Weiss MG, Nielsen PH, James S, Thelin S, Modrau IS. Clinical Outcomes After Surgical Revascularization Using No-Touch Versus Conventional Saphenous Vein Grafts: Mid-Term Follow-Up of Propensity Score Matched Cohorts. Semin Thorac Cardiovasc Surg. 2023 Summer;35(2):228-236. doi: 10.1053/j.semtcvs.2021.12.002. Epub 2021 Dec 5. PMID 34879223

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT06496321/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT06496321/ICF_001.pdf